CLINICAL TRIAL: NCT05487963
Title: Tolerability and Effectiveness of CGB 500 Topical Ointment, 1% Tofacitinib, for the Treatment of Atopic Dermatitis: a Randomized, Double-Blind, Vehicle-Controlled Study
Brief Title: Tolerability and Effectiveness of CGB-500 Topical Ointment, 1% Tofacitinib, for the Treatment of Atopic Dermatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CAGE Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CGB-500-001
Record Dates: First submitted 2022-08-01; First posted 2022-08-04 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-05

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CGB-500 topical ointment, 1% tofacitinib (Experimental)
  Interventions: Drug: Tofacitinib Citrate
- Vehicle topical ointment (Placebo Comparator)
  Interventions: Other: placebo ointment

INTERVENTIONS:
Drug: Tofacitinib Citrate — Topical application of a pea-sized amount of ointment (active or vehicle) over a maximum surface of 30 cm2 up to 2 times a day.
  Arms: CGB-500 topical ointment, 1% tofacitinib
Other: placebo ointment — Topical application of a pea-sized amount of ointment (active or vehicle) over a maximum surface of 30 cm2 up to 2 times a day.
  Arms: Vehicle topical ointment

SUMMARY:
The objective of the proposed study is to evaluate the tolerability and effectiveness of a 1% topical ointment of tofacitinib for the treatment of mild to moderate atopic dermatitis in adults. Adult patients with a diagnosis of atopic dermatitis for at least 6 months will be treated with the test product or placebo for a period of 8 weeks with a follow-up visit at 12 weeks. The primary endpoints are safety and tolerability of CGB-500 Ointment and a comparison of effectiveness of CGB-500 Ointment and Vehicle Ointments in treating lesion(s) of mild to moderate atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient, male or female of any race, 18 years of age or older. Female subjects of childbearing potential must have a negative urine pregnancy test at Baseline and practice a reliable method of contraception throughout the study.
2. Have a clinical diagnosis of atopic dermatitis for at least 6 months prior to Day 0 (at the Screening and Baseline visit) that has been clinically stable for ≥3 months prior to dose administration and is confirmed to be atopic dermatitis according to the criteria of Hanifin and Rajka.
3. Have an IGA score of 2 (mild) or 3 (moderate) at Day 0.
4. Have an EASI score of 1.1 to 12.0 (i.e., mild or moderate).
5. Have atopic dermatitis on the arms and other body parts covering at least 2% of total BSA and up to and including 12% of total Body Surface Area (BSA) at Day 0.
6. Have a presence of 1 to 3 target atopic dermatitis lesions of total surface area of 15 to 30 cm2, located on the body part visible to the subject. This is the target lesion(s) that will be treated in this study.
7. Agree to use only low potency corticosteroid (up to 1% hydrocortisone) topical cream or ointment for the other affected parts of the body that are not being treated with the investigational product in the study, and at least 5 cm away from the treated area.
8. In general, good health as determined by medical history and physical examination at the time of screening (Investigator discretion).
9. Have a Peak Pruritus NRS score of ≥30 on the of scale 0 to 100, especially on the target lesions.
10. Ability to follow study instructions and likely to complete all required visits.
11. Have signed the Institutional Review Board (IRB)-approved Informed Consent Form (ICF) prior to any study-related procedures being performed.
12. Participating in any other clinical trial from 30 days prior to Screening and throughout the planned 12-week study period.

Exclusion Criteria:

1. Female subjects who are pregnant, breast-feeding, or of childbearing potential and not practicing reliable birth control.
2. Known hypersensitivity or previous allergic reaction to any constituent of the Investigational Product (i.e., essential oils, choline, phosphatidylcholine, glycerol, propylene glycol, polyethylene glycol).
3. Any transient flushing syndrome.
4. Severe atopic dermatitis.
5. Unstable course of atopic dermatitis (spontaneous improvement over time).
6. Skin infections (bacterial, fungal or viral) that can interfere with reliable atopic dermatitis assessments.
7. Basal cell carcinoma within 6 months of Baseline (Visit 1).
8. History of confounding skin conditions, e.g., psoriasis, rosacea, erythroderma, or ichthyosis or presence of Netherton's syndrome, immunological deficiencies or diseases, HIV, diabetes, malignancy, serious active or recurrent infection, clinically significant severe renal insufficiency, or severe hepatic disorders.
9. Use within 1 month prior to Baseline of 1) oral or intravenous corticosteroids, 2) UVA/UVB therapy, 3) PUVA (Psoralen plus UltraViolet A) therapy, 4) tanning booths, 5) non-prescription UV light sources, 6) immunomodulators or immunosuppressive therapies, 7) interferon, 8) cytotoxic drugs, 9) crisaborole, 10) pimecrolimus, or 11) injectable biologics (e.g. Dupixent).
10. Use within 14 days of Baseline of: 1) systemic antibiotics, 2) systemic JAnus Kinase (JAK) products, 3) calcipotriene or other vitamin D preparations, or 4) retinoids.
11. Use within 7 days prior to Baseline of: 1) antihistamines, 2) topical antibiotics, 3) topical corticosteroids or 4) other topical drug products.
12. Use within 24 hours prior to Baseline of any topical product (e.g., sunscreens, lotions, creams, emollients, moisturizers) in the areas to be treated.
13. Known allergy or hypersensitivity to tofacitinib or any other component of the Investigational Product (i.e., essential oils, choline, phosphatidylcholine, glycerol, propylene glycol, polyethylene glycol).
14. Uncontrolled systemic disease.
15. Foreseen unprotected and intense/excessive UV exposure during the study.
16. Scheduled or planned surgical procedures during the study.
17. Unable or unwilling to comply with any of the study requirements.
18. Medical or psychiatric conditions, or a personal situation, that may increase the risk associated with study participation or may interfere with interpretation of study results or subject compliance and, in the opinion of the Principal Investigator, makes the subject inappropriate for study entry.
19. Clinically significant alcohol or drug abuse, or history of poor cooperation or unreliability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | 8 weeks
  Frequency of subjects with Treatment-Emergent Adverse Events (TEAEs).
  • Frequency of subjects with skin irritation TEAEs and any other adverse skin reactions.
Effectiveness | 8 weeks
  Percent change from baseline in lesional Eczema Area and Severity Index (EASI) score at Week 8. EASI is scored on a 0 - 6 scale with 0 being no eczema and 6 being 100% of the area affected by eczema.

SECONDARY OUTCOMES:
Investigator's Global Assessment (IGA) | 8 weeks
  Percentage of subjects achieving Investigator's Global Assessment (IGA) response of 'Clear' (Score 0) or 'Almost Clear' (Score 1) at Week 8.
Eczema Area and Severity Index (EASI) | 8 weeks
  Percentage of subjects who achieve a ≥75% improvement from baseline in lesional EASI score at Week 8
Pruritis | 8 weeks
  Change from baseline in peak lesional pruritus (itching) Numeric Rating Scale (NRS) score at Week 8. NRS goes from 0 to 10; with 0 signifying no itching and 10 signifying worst itch imaginable.

CONTACTS AND LOCATIONS:
Locations (1):
- Kani Clinic, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: No